CLINICAL TRIAL: NCT07080658
Title: A Phase I Study to Investigate The Mass Balance and Biotransformation of WPV01 in Healthy Adult Chinese Male Participants
Brief Title: [14C] Study to Investigate the Mass Balance and Biotransformation of WPV01 in Healthy Adult Chinese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Westlake Pharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WPV01-MB-01
Record Dates: First submitted 2024-07-12; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- WPV01 (Experimental)
  Interventions: Drug: [14C]-WPV01

INTERVENTIONS:
Drug: [14C]-WPV01 — Single oral dose of 600 mg [14C]-WPV01

SUMMARY:
This is a single-center, non-randomized, open-label, single-dose, Phase I clinical study to evaluate the mass balance and biotransformation, safety and tolerability of WPV01 in healthy adult chinese male participants following a single oral administration of [14C] WPV01.

DETAILED DESCRIPTION:
This trial is planned to enroll 6-8 healthy Chinese male subjects. Each subject is administered a single oral dose containing 600 mg/approximately 100 µCi [14C]WPV01 suspension on the first day of the trial in fasting condition.

Whole blood, plasma, urine and fecal samples are collected at defined time points/periods during the test. The whole blood/plasma partition ratio, pharmacokinetic parameters of total radioactivity in plasma, recovery and excretion pathway data of [14C]WPV01 are calculated by measuring the total radioactivity. The major metabolic elimination pathways and characterization of WPV01 in the human body, as well as circulating metabolites that are close to or above 10% of total plasma radioactivity exposure, are obaitned from structural characterization of plasma, urine and fecal radio-metabolite profiles and major metabolites.

All excreted urine and fecal samples are collected at specified time intervals from 0 to 336h post-dose and and blood samples are collected at specified time points from 0 to 144h post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males
* Participants aged ≥18 years and ≤55 years old
* Body weight: Body mass index (BMI) between 19.0 and 26.0 kg/m2 (including borderline values), body weight no less than 50.0 kg.
* Voluntarily participate in the clinical trial and sign the informed consent
* Able to communicate well with the investigator and able to complete the trial in accordance with the protocol

Exclusion Criteria:

* Participants who have abnormalities and clinical significance after comprehensive physical examination, vital signs, routine laboratory tests, thyroid function, chest CT, abdominal ultrasound, etc.
* Participants whose 12-lead electrocardiogram test results show corrected QT interval ≥450 msec
* Participants who is positive for Hepatitis B Surface Antigen, Hepatitis C Antibody, HIV Antibody and Syphilis Antibody
* Participants who have used any drug that inhibits or induces hepatic drug metabolizing enzymes within 30 days prior to the screening period
* Participants who have used any prescription medication, over-the-counter medication, herbal or dietary supplements, such as vitamins, calcium supplements, within 14 days prior to the screening period
* Participants who have a history of any clinically serious disease or disease/condition that, in the opinion of the investigator, may affect the results of the test, including, but not limited to, a history of circulatory, respiratory, endocrine, neurological, gastrointestinal, urological, or hematological, immunological, psychiatric, and metabolic disorders
* Participants who have any condition that may affect drug absorption, e.g., gastrectomy, cholecystectomy, gastric bypass, duodenotomy, colectomy, history of inflammatory bowel disease
* Participants who have history of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, ventricular tachycardia, atrioventricular block, QT prolongation syndrome, or symptoms of QT prolongation syndrome, and a family history of the disease (as evidenced by genetic predisposition or by the death of a close family member from a cardiac cause at a young age).
* Participants who have undergone major surgery within 6 months prior to the screening period or whose surgical incisions have not completely healed; major surgery includes, but is not limited to, any surgery with significant risk of hemorrhage, prolonged general anesthesia, or incisional biopsy or significant traumatic injury
* Participants who have specific allergic history, such as those with a known history of allergy to two or more substances; or those who, in the judgment of the investigator, may be allergic to the test drug or its excipients
* Participants who have perianal disease with regular/ongoing blood in stool, irritable bowel syndrome, inflammatory bowel disease
* Participants who have habitual constipation or diarrhea
* Participants who are alcohol abusers or regularly drink alcohol in the 6 months prior to the screening period, i.e., more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits at 40% alcohol by volume or 150 mL of wine); or an alcohol breath test result of >0 mg/dL at the time of the screening period
* Participants who smoked >5 cigarettes per day in the 3 months prior to the screening period or habitually used nicotine-containing products and were unable to quit during the trial period
* Participants who are substance abusers or use soft drugs (e.g., marijuana) in the 3 months prior to the screening period or use of hard drugs (e.g., cocaine, amphetamines, phenylcyclohexylpiperidine, etc.) in the 1 year prior to the screening period; or a positive urine drug test at the screening period
* Participants who consume grapefruit juice or excessive amounts of tea, coffee and/or caffeinated beverages that cannot be stopped during the trial period
* Participants who are exposed to radiation for prolonged periods of time; or who have had significant radiation exposure (≥2 chest/abdominal CTs, or ≥3 other types of X-rays) or participated in radiopharmaceutical labeling tests within 1 year prior to testing
* Participants who are with a history of needle and blood sickness, those who have difficulty in blood collection or cannot tolerate venipuncture blood collection
* Participation in any other clinical trial (including clinical trials such as drugs and devices) within 3 months prior to the screening period
* Participants who have vaccinated within 1 month prior to screening or scheduled to be vaccinated during the trial period
* Participants who plan to have children or donate sperm during the trial and within 1 year after completion of the trial, or who do not agree that the subject and his/her spouse should use strict contraception during the trial and within 1 year after completion of the trial
* Participants who have had blood loss or donated up to 400 mL of blood within 3 months prior to the screening period, or those who have received a blood transfusion within 1 month
* Participants who, in the opinion of the investigator, have any factors that make participation in this trial inappropriate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adult males
Enrollment: 6 (Actual)
Dates: Start 2023-07-23 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Total recovery and cumulative recovery of total WPV01-related radioactive material in excreta (urine and feces) | Up to 168 hours(approx) from drug administration
Total radioactivity of WPV01-related substances in human plasma | Up to 168 hours(approx) from drug administration
Ratio of total WPV01-related radioactivity concentrations in human whole blood and plasma at different time points | Up to 168 hours(approx) from drug administration
WPV01 and its metabolites in human plasma as a percentage of total plasma radioactivity exposure | Up to 168 hours(approx) from drug administration
WPV01 and its metabolites in human excreta (urine and feces) as a percentage of total urine/feces radioactivity exposure | Up to 168 hours(approx) from drug administration
Identification of metabolites in plasma | Up to 168 hours(approx) from drug administration
Identification of metabolites in urine | Up to 168 hours(approx) from drug administration
Identification of metabolites in feces | Up to 168 hours(approx) from drug administration

SECONDARY OUTCOMES:
Time to maximum plasma concentration of WPV01 and its metabolites (if applicable) in plasma | Up to 168 hours(approx) from drug administration
Maximum plasma concentration of WPV01 and its metabolites (if applicable) in plasma | Up to 168 hours(approx) from drug administration
Terminal half-life of WPV01 and its metabolites (if applicable) in plasma | Up to 168 hours(approx) from drug administration
Number of Participants With Adverse Events | At least up to 14 days from drug administration
Area under the plasma concentration-time curve of WPV01 and its metabolites (if applicable) in plasma | Up to 168 hours(approx) from drug administration
Mean residence time of WPV01 and its metabolites (if applicable) in plasma | Up to 168 hours(approx) from drug administration
Number of Participants With Clinically Notable Vital Signs | At least up to 14 days from drug administration
Number of Participants With Clinically Notable Laboratory Tests | At least up to 14 days from drug administration
Number of Participants With Clinically Notable ECG Tests | At least up to 14 days from drug administration
Number of Participants With Clinically Notable Physical Examination | At least up to 14 days from drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No